CLINICAL TRIAL: NCT04522557
Title: Type I Interferon Alfa-2a in Postmastectomy Breast Reconstruction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Shicheng Su, Director of Shuhua Breast Cancer Research Center of Sun Yat- sen Memorial Hospital, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2020-KY-051
Record Dates: First submitted 2020-08-18; First posted 2020-08-21 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Breast Neoplasms
Keywords: Breast reconstruction; Implants; Interferon (IFN)
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Participants with breast cancer enrolled in grou (Experimental)
  Interventions: Drug: IFNα-2a

INTERVENTIONS:
Drug: IFNα-2a — After mastectomy, it is used in the cavity of breast before conducting implantation.

SUMMARY:
RATIONALE: Implant-based reconstruction have become the most popular choices of reconstruction for women undergoing breast mastectomy. Postoperative complications like infection and tumor recurrence limit its application. Interferons (IFNs) are pleiotropic cytokines that involve in immunoregulatory, anticancer and restricting infection. Especially, type I IFN signaling is reported favourable for the success of conventional chemotherapeutics, radiotherapy and immunotherapy. In addition, type I IFN can regulate the activity of almost all immune cell types (including T cells, macrophages and innate lymphocytes), creating a well-established immune environment to defense infectious and relapsing disease. Implants are rapidly coated with extracellular matrix proteins and immune protein components for the formation of a typical capsule. At the specific time point before implantation, the locally utilized of IFN in intracavity breast is assumed to modify cellular immune responses thus contributing to decreasing infection and tumor recurrence.

PURPOSE: This non-randomized phase I trial aims to explore dose range of IFNα-2a. Adverse events are observed to assess drug safety and human tolerance index.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the informed consent.
2. Female aged between 18 and 70 years.
3. Pathologically diagnosed operable breast cancer.
4. WHO Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
5. Newly diagnosed breast cancer.
6. The important organ functions meet the following criteria:

   * WBC >=3.0 x 10^9/L; Neutrophilic granulocytes >=1.5×10^9/L; Platelet >=100 x 10^9/L; Hb >=9 g/dL;
   * Total bilirubin no more than 1.5 times the normal upper limit (ULN); AST and ALT no more than 1.5 times ULN; AKP no more than 2.5 times ULN;
   * Serum creatinine no more than 1.5 times ULN or Clearance rate of creatinine >= 60ml/min;
   * Thyroid stimulating hormone (TSH) <= ULN (T3, T4 levels need to be detected simultaneously if abnormalities, the patient can be included if T3, T4 levels is normal);
   * LVEF basement >= 50%.

Exclusion Criteria:

1. Evidence of distant metastasis.
2. Any contraindication of nipple-areolar complex (NAC) saving mastectomy (NSM):

   * Intraoperative biopsy revealed carcinoma invasion of NAC.
   * Paget's disease of breast.
   * Tumor distant from NAC less than 1 cm.
3. Any invasive malignancy diagnosed within previous 5 years (other than successfully treated cervical carcinoma in situ, skin basal cell carcinoma or cutaneous squamous cell carcinoma).
4. At least 4 months since prior interferon therapy.
5. At least 3 weeks since prior major surgery requiring general anesthesia.
6. At least 3 weeks since prior radiotherapy or chemotherapy.
7. Hypersensitivity to interferon or other components: urticaria, angioedema, bronchial stenosis, anaphylaxis, or Stevens-Johnson syndrome.
8. Prior organ allograft.
9. Use of an unlicensed or other investigational drug within 4 weeks.
10. Any severe comorbidities, inability to give informed consent or unavailability for follow-up, including but not limited to any of the following:

    * Heart failure above NYHA class 2 level; high-risk uncontrollable arrhythmia; unstable angina pectoris; myocardial infarction within 1 intervention.
    * Chronic obstructive pulmonary disease requires treatment.
    * Chronic liver disease (cirrhosis, chronic active hepatitis, etc.).
    * Cerebrovascular accident occurred within 6 months.
    * Severe epilepsy or central nervous system diseases.
    * Hypertension which cannot be well controlled by antihypertensive drugs.
    * Abnormal coagulation, bleeding tendency, or receiving thrombolysis or anticoagulant therapy.
    * Chronic renal insufficiency.
    * Active infection.
    * Psychiatric disability, etc.
11. Pregnant or lactating women.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-07-14 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 7 days after surgery
  Dose-limiting toxicity (DLT), defined as certain grade II toxicity such as nephrotoxicity and cardiotoxicity, grade III non-hematologic toxicity and grade IV hematologic toxicity.
Maximal tolerable dose (MTD) | 7 days after surgery
  Maximal tolerable dose (MTD), defined as a dose level where 2 or more subjects among 6 subjects suffering DLT. If the experiment reached the set maximum dose without any DLT occurring, the maximum dose was defined as MTD.

SECONDARY OUTCOMES:
Adverse events (AE) | 7 days after surgery
Server adverse events (SAE) | 7 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Shicheng Su, M.D.,Ph.D., Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Shicheng Su, Guangzhou, Guangdong, China